CLINICAL TRIAL: NCT06446999
Title: The Effect of Yoga-Based Breathing Exercise on Pain, Fatigue, Insomnia, and Self-Efficacy in Individuals Undergoing Colorectal Cancer Surgery-Randomized Controlled Study
Brief Title: Yoga-Based Breathing Exercise, Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayFG
Record Dates: First submitted 2024-05-11; First posted 2024-06-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-07

CONDITIONS: Symptoms and Signs
Keywords: Colorectal cancer surgery; Yoga-Based Breathing Exercise; Pain; Fatigue; İnsomnia; Self Efficacy
MeSH Terms: conditions — Signs and Symptoms; Pain; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 1. Experimental group: A protocol containing yoga-based breathing exercises will be used. The audio recording of this breathing exercise protocol will be uploaded to the video. After verbal information is given about how to do the exercise, the patient will be listened to the audio recording video and will be explained how to do it in practice. Then, the patient will be placed in a comfortable position by wearing headphones and will be allowed to exercise. The patient will be asked to do yoga-based exercise twice a day, the night before the surgery, once in the morning and once in the evening before going to bed for 3 days after the surgery.
  2. Control group: Continuity of routine treatment and care of the patients included in the control group will be ensured.
Who Masked: Outcomes Assessor
Masking Description: The data obtained as a result of the research will be coded as 'A' and 'B' by the researcher and transferred to the computer. In order to prevent bias in the evaluation of the data, the analysis of the coded data will be carried out by an independent statistician, thus ensuring statistician blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-Based Breathing Exercise (Experimental): A protocol containing yoga-based breathing exercises will be used. The audio recording of this breathing exercise protocol will be uploaded to the video. After verbal information is given about how to do the exercise, the patient will be listened to the audio recording video and will be explained how to do it in practice. Then, the patient will be placed in a comfortable position by wearing headphones and will be allowed to exercise. The patient will be asked to do yoga-based exercise twice a day, the night before the surgery, once in the morning and once in the evening before going to bed for 3 days after the surgery.
  Interventions: Other: Yoga-Based Breathing Exercise
- Control (No Intervention): Continuity of routine treatment and care of the patients included in the control group will be ensured.

INTERVENTIONS:
Other: Yoga-Based Breathing Exercise — Breathing Exercise Protocol Purpose: This protocol is a guide prepared for patients who agree to participate in the study within the scope of scientific research to do breathing exercises.
  Materials Required: A comfortable chair/a comfortable bed to lie on and comfortable clothing.
  Exercise Duration: Approximately 20 minutes Exercise Time and Frequency: It should be done twice a day, at the same time, in the morning and in the evening.
  You can do the exercise before going for a walk in the corridor in the morning and before going to sleep in the evening.
  Normal Breathing and Focusing on Breathing (3 minutes) Alternate Nose Breathing-Nadi Shodhana (15-20 times/6 minutes) Normal Breathing and Focusing on Breathing (3 minutes) Bhramari Pranayama-Bee Buzzing Sound(8-10 times/5 minutes) Normal Breathing and Focusing on Breathing (3 minutes)
  Arms: Yoga-Based Breathing Exercise

SUMMARY:
This study was designed as a prospective, parallel two groups and randomized controlled study with an experimental-control group to evaluate the effect of yoga-based breathing exercise on pain, fatigue, insomnia and self-efficacy in individuals undergoing colorectal cancer surgery. The sample size of the study was conducted with 60 patients, 30 in the control group and 30 in the experimental group, according to the results of a similar study with the G*Power 3.1., 9.7 program, with α = 0.05, 80% power and 0.648 effect, and taking into account possible losses. was planned. Research inclusion criteria; Patients who underwent colorectal cancer surgery for the first time were those who were 18 years of age or older, had a mobile phone suitable for downloading the yoga-based breathing exercise video, used the same type and dose of painkillers, and volunteered to participate in the study. "Personal Information Form", "VAS Pain Scale", "Brief Fatigue Inventory", "Richard Campbell Sleep Scale" and "Health Promotion Strategies Used by Patients Scale" will be used to collect data. Participants assigned to the experimental group will be provided with breathing exercises using a protocol containing Yoga-based breathing exercises. In order to conduct the research, approval will be obtained from KTO Karatay University Non-Drug and Medical Device Research Ethics Committee, ethics committee approval and permission will be obtained from the institution where the research will be conducted. Participation in the study is voluntary and written consent will be obtained from the participants. The data will be evaluated in the IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA) statistical package program. A level of p<0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Colorectal cancers are the third most common type of cancer in terms of incidence worldwide and the second leading cause of death. Surgical treatment, chemotherapy and radiotherapy are generally used in the treatment of colorectal cancers. Side effects such as pain, nausea-vomiting, intestinal problems, and fatigue may occur after colorectal cancer surgery (CRCS). In addition, in patients who subsequently receive chemotherapy or radiotherapy, these patients may experience symptom distress and their quality of life may be negatively affected due to side effects such as nausea, vomiting, diarrhea, malnutrition, peripheral neuropathy and fear of cancer recurrence. Pharmacological methods in the management of fatigue are quite limited, and the effect of non-pharmacological approaches such as cognitive behavioral therapies, relaxation, exercise, training of patients and their relatives for fatigue management, exercise, cognitive behavioral therapies, and meditation is effective. Studies evaluating it are increasing. However, it has been stated that very few (10%) of cancer patients experiencing severe fatigue do yoga to manage fatigue. This research was planned to evaluate the effect of yoga-based breathing exercise on pain, fatigue, insomnia and self-efficacy in individuals undergoing colorectal cancer surgery.

Type of Research: This study was designed as a prospective, parallel 3-group and randomized controlled study with an experimental-control group to evaluate the effect of yoga-based breathing exercise on pain, fatigue, insomnia and self-efficacy in individuals undergoing colorectal cancer surgery.

Place and Time of the Research: The research will be conducted at Necmettin Erbakan University Meram Medical Faculty General Surgery Clinic between 01 September 2023 and 30 July 2024.

Population and Sample of the Research: The research population will consist of patients who come for colorectal cancer surgery between 01 September 2023 and 30 July 2024 at Necmettin Erbakan University Meram Faculty of Medicine General Surgery Clinic, where the research will be conducted. The sample number of the study was determined according to the results of a similar study with the G*Power 3.1., 9.7 program with α = 0.05 and 80% power and 0.648 effect. The sample was determined as 50 patients, 25 patients in the experimental group and 25 patients in the control group. Considering possible losses during the study, it was planned to include a total of 60 patients, 30 patients in the experimental group and 30 patients in the control group.

Data Collection Tools: "Personal Information Form", "VAS Pain Scale", "Brief Fatigue Inventory", "Richard Campbell Sleep Scale" and "Health Promotion Strategies Used by Patients Scale" will be used to collect data.

VAS Pain Scale: It is a scale used to evaluate pain by giving a value between 0 and 10. A score of 0 means no pain, and a score of 10 means unbearable pain. As the score increases, the severity of pain increases.

Brief Fatigue Inventory: The scale evaluates the level of fatigue in the last 24 hours and the reflection of this fatigue on activities in daily life (general activity, mood, walking ability, work life, relationships with other people, joy of life). KYE; It consists of a total of 9 items, 3 items assessing fatigue, general fatigue, and 6 items assessing the impact of fatigue on daily life. Individuals score all items between "0" (no fatigue at all) and "10" (the most severe fatigue you can experience), taking into account the last 24 hours.

Richard Campbell Sleep Scale: The scale developed to determine sleep quality consists of six items: depth of night sleep, time to fall asleep, frequency of waking up, time to fall asleep when woken up, quality of sleep and noise level in the environment. Visual analog scale technique was applied for all expressions. RCUÖ average value; Scale variables are calculated by adding the mean scores and dividing by five. There is only a total score in the scale and the evaluation is made on the average of this score. A total score of the scale between 0 and 25 indicates poor sleep, and a score between 76 and 100 indicates good sleep. An increase in the total score average defines a positive increase in sleep quality.

Health Promotion Strategies Used by Patients Scale: The health promotion strategies used by patients scale was developed. This scale is a 29-item self-report scale. The scale, which initially consisted of 36 items and 4 subscales, was rearranged in 2001. With the factor analysis study called "Confirmatory Factor Analysis", the number of scale items was reduced to 29 and 3 sub-dimensions were defined. These sub-dimensions are: coping with stress, decision making and positive behavior. 1st to 10th of the scale. item, coping with stress sub-dimension, 11th-13th. items decision-making sub-dimension, 14th-29th. The items are the positive behavior subdimension.

Implementation of the Research: Patients who will undergo CRC will be given verbal information about the research before surgery, and those who agree to participate in the research will be evaluated for compliance with the inclusion criteria. The purpose of the research and how it will be implemented will be explained to the patient who meets the criteria for inclusion in the research, and their written consent will be obtained. Initial assessments will be made regarding sociodemographic and health history, VAS Pain score, Fatigue, Insomnia and Self-Efficacy level before surgery/pre-intervention. After the initial evaluation, patients will be assigned according to randomization. For the second evaluation, the VAS Pain score, Fatigue, Insomnia and Self-Efficacy levels of the control and experimental groups will be evaluated on the 4th day after surgery.

Experimental group: A protocol containing yoga-based breathing exercises will be used. The audio recording of this breathing exercise protocol will be uploaded to the video. After verbal information is given about how to do the exercise, the patient will be listened to the audio recording video and will be explained how to do it in practice. Then, the patient will be placed in a comfortable position by wearing headphones and will be allowed to exercise. The patient will be asked to do yoga-based exercise twice a day, the night before the surgery, once in the morning and once in the evening before going to bed for 3 days after the surgery.

Control group: Continuity of routine treatment and care of the patients included in the control group will be ensured. The control group will be recruited before preoperative assignment to patients. After the final test of the patients, information will be given about breathing exercises, and patients who want to do breathing exercises will be provided with a video link uploaded to their mobile phones.

Ethical Dimension of the Research: In order to conduct the research, ethics committee approval was obtained from KTO Karatay University Non-Pharmaceutical and Non-Medical Device Research Ethics Committee and permission was obtained from the institution where the research will be conducted. Participation in the study is voluntary and written consent will be obtained from the participants. To avoid bias, Clinical Trials protocol registration will be made after obtaining permission from the ethics committee.

Statistical Evaluation of Research Data: The data will be evaluated in the IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA) statistical package program. Descriptive statistics will be given as number of units (n), percentage (%), mean ± standard deviation, median (M), minimum (min) and maximum (max) values. The normal distribution of the data of numerical variables will be evaluated with the Shapiro Wilk normality test. Homogeneity of variances will be evaluated with the Levene test. To evaluate the differences between two independent groups, "Student's t Test" is used when parametric test prerequisites are met; When this could not be achieved, the "Mann Whitney-U test" was used. A level of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Having colo-rectal surgery for the first time
* Have a mobile phone suitable for downloading the yoga-based breathing exercise video,
* Use the same type and dose of painkillers,
* No communication barrier
* Volunteer to participate in the study.

Exclusion Criteria:

* Using sleeping pills,
* Having a physical disability in doing breathing exercises,
* Being diagnosed with a psychiatric disease,
* Having been doing yoga breathing exercises for the last six month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) - Pain Scale | One minute
  A 10 cm ruler has been designed with painlessness on one side and the most severe pain possible on the other side. This ruler is known as the Visual Analog Scale (VAS) for visual comparison. In the evaluation of the scale, "0" indicates no pain, "1-3" indicates mild pain, "4-6" indicates moderate pain, and "7-10" indicates severe pain levels.
Brief Fatigue Inventory | Two minutes
  In the evaluation of fatigue, 0 points; no fatigue, 1-3 points; low fatigue, 4-6 points moderate fatigue, 7-9 points; extreme fatigue, 10 points; Fatigue is rated at the highest level.
Richard Campbell Sleep Scale | Two minutes
  It is a scale consisting of 6 items that assess the depth of nighttime sleep, the time it takes to fall asleep, the frequency of awakenings, the duration of wakefulness upon awakening, the quality of sleep, and the level of noise in the environment. Scores on the scale range from "0-25" indicating very poor sleep to "76-100" indicating very good sleep. While evaluating the total score of the scale based on 5 items, the 6th item, which assesses the level of noise in the environment, is excluded from the total score assessment. As the score on the scale increases, the quality of patients' sleep also increases.
A measure of self-care self-efficacy | Two minutes
  The minimum score obtained from the scale is 29 and the maximum score is 145. An increase in score indicates that the level of self-efficacy regarding self-care behaviors has increased.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gündogdu, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared when necessary.

REFERENCES:
- [Background] Ban KA, Gibbons MM, Ko CY, Wick EC, Cannesson M, Scott MJ, Grant MC, Wu CL. Evidence Review Conducted for the Agency for Healthcare Research and Quality Safety Program for Improving Surgical Care and Recovery: Focus on Anesthesiology for Colorectal Surgery. Anesth Analg. 2019 May;128(5):879-889. doi: 10.1213/ANE.0000000000003366. PMID 29649026
- [Background] Jaya P, Thakur A. Effect of Progressive Muscle Relaxation Therapy on Fatigue and Psychological Distress of Cancer Patients during Radiotherapy: A Randomized Controlled Trial. Indian J Palliat Care. 2020 Oct-Dec;26(4):428-432. doi: 10.4103/IJPC.IJPC_236_19. Epub 2020 Nov 19. PMID 33623302
- [Background] Kirca K, Kutluturkan S. The effect of progressive relaxation exercises on treatment-related symptoms and self-efficacy in patients with lung cancer receiving chemotherapy. Complement Ther Clin Pract. 2021 Nov;45:101488. doi: 10.1016/j.ctcp.2021.101488. Epub 2021 Oct 2. PMID 34619419
- [Background] Lev EL, Owen SV. A measure of self-care self-efficacy. Res Nurs Health. 1996 Oct;19(5):421-9. doi: 10.1002/(SICI)1098-240X(199610)19:53.0.CO;2-S. PMID 8848626
- [Background] Scheepers ERM, Vink GR, Schiphorst AHW, Emmelot-Vonk MH, van Huis-Tanja LH, Hamakerl ME. Health-related quality-of-life trajectories during/after surgery and adjuvant chemotherapy in patients with colon cancer. Eur Geriatr Med. 2023 Jun;14(3):565-572. doi: 10.1007/s41999-023-00750-9. Epub 2023 Mar 25. PMID 36964869
- [Background] Schmidt ME, Bergbold S, Hermann S, Steindorf K. Knowledge, perceptions, and management of cancer-related fatigue: the patients' perspective. Support Care Cancer. 2021 Apr;29(4):2063-2071. doi: 10.1007/s00520-020-05686-5. Epub 2020 Aug 29. PMID 32860177
- [Background] Yin L, Fan L, Tan R, Yang G, Jiang F, Zhang C, Ma J, Yan Y, Zou Y, Zhang Y, Wang Y, Zhang G. Bowel symptoms and self-care strategies of survivors in the process of restoration after low anterior resection of rectal cancer. BMC Surg. 2018 Jun 4;18(1):35. doi: 10.1186/s12893-018-0368-5. PMID 29866087
- [Result] Akin S, Can G, Durna Z, Aydiner A. The quality of life and self-efficacy of Turkish breast cancer patients undergoing chemotherapy. Eur J Oncol Nurs. 2008 Dec;12(5):449-56. doi: 10.1016/j.ejon.2008.07.006. Epub 2008 Oct 7. PMID 18842460